CLINICAL TRIAL: NCT07035327
Title: Effect of the Resistance-cognitive Dual-task Training on Frailty Status and Cognitive Function in Frail Community-dwelling Older Adults With Chronic Musculoskeletal Pain: A Pilot Randomized Controlled Trial
Brief Title: Dual-task Training for Frail Older Adults With Chronic Musculoskeletal Pain (Pilot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, YAU King Wai Derek, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20250310005
Record Dates: First submitted 2025-06-05; First posted 2025-06-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Chronic Musculoskeletal Pain; Frailty
Keywords: Chronic musculoskeletal pain; Frailty; Dual-task training; Pain management
MeSH Terms: conditions — Frailty; Agnosia | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomization and group assignment will be performed by an investigator not involved in recruitment or assessment. After participants' eligibility for enrolment is confirmed, a researcher will use a computer to automatically generate a random sequence using Excel software (Microsoft Corporation, Redmond, USA) to generate random integers, with odd numbers being the experimental group and even numbers being the control group. The grouping information will be stored in a separate folder. Participants will undergo the corresponding exercise program which will be supervised by the researcher. The outcome assessor will be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group - Dual-task training program (Experimental): Participants in the intervention group will engage in a dual-task training program, in which resistance training will be incorporated with cognitive tasks (2 sessions per week for 10 weeks consecutively). The training sessions will take place in an academic institution under the guidance and supervision from the members of research team.
  Interventions: Other: Dual-task training program
- Control group - Resistance exercise (Active Comparator): Subjects in the control group will perform the resistance exercises only (2 sessions per week for 10 weeks consecutively) without receiving any cognitive training. The training sessions will take place in an academic institution under the guidance and supervision from the members of our research team.
  Interventions: Other: Resistance exercise

INTERVENTIONS:
Other: Dual-task training program — Participants in the intervention group will engage in a dual-task training program, in which resistance training will be incorporated with cognitive tasks.
  - Resistance training: Participants will be instructed to perform the following exercises with proper form: (1) squat to chair, (2) seated unilateral hip flexion, (3) seated unilateral knee extension, (4) standing unilateral knee flexion and (5) bilateral calf raise. The lower limb exercises will be followed by four upper limb exercises: (6) seated elbow flexion, (7) twisting a towel, (8) seated horizontal opening of arms and elbow, (9) seated diagonal opening of arm and elbow.
  - Cognitive task: Subjects will be asked to perform a verbal fluency task or mental arithmetic tasks simultaneously with the resistance training exercises.
  Arms: Intervention group - Dual-task training program
Other: Resistance exercise — Subjects in the control group will perform the resistance exercises only without receiving any cognitive training. Ten-minute warm-up and cool-down sessions will precede and follow each exercise session.
  Arms: Control group - Resistance exercise

SUMMARY:
The goal of this clinical trial is to investigate the feasibility and effect of a 10-week dual-task training program on frailty status in community-dwelling older adults with frailty and chronic musculoskeletal pain.

Main question: Is a 10-week dual-task training program, that combines resistance and cognitive training, feasible and accepted by community-dwelling older adults who have frailty and chronic musculoskeletal pain, and what is the effect of a 10-week dual-task training program on the frailty status in community-dwelling older adults who have frailty and chronic musculoskeletal pain?

Participants will attend supervised training sessions (either dual-task training [Intervention group] or resistance exercise [Control group]) for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults, of either sex, aged 60 years or above,
* living in Hong Kong, being able to read and communicate verbally,
* screened frail using the Tilburg Frailty Indicator (TFI) (total score ≥5) with report of memory problems (question 9) (Gobbens et al., 2010),
* experiencing any CMP with a pain level higher or equal to 4 in the numerical pain rating scale over a consecutive 3-month period.

Exclusion Criteria:

Any individuals with either of the following will be excluded:

* absence of frailty,
* surgical procedure in the lower limbs or the vertebral column;
* wheelchair bound or inability to walk for five minutes;
* severe balance impairment;
* uncompensated cardiac or vascular condition;
* acute inflammatory musculoskeletal conditions;
* ongoing cancer; dementia;
* neurological diseases such as stroke, Parkinson's disease, cerebellar disease, myelopathy, and peripheral neuropathy;
* mental illnesses such as schizophrenia, bipolar, psychosis, borderline personality disorder;
* illiteracy.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability | Post-treatment (Week 10)
  The primary outcomes will be feasibility and acceptability of the dual task training program. Feasibility will be evaluated through recruitment and compliance rates of the program. Recruitment rate will be defined as the total number of participants recruited out of the total number of participants screened. Treatment compliance will be defined as the proportion of scheduled sessions attended in each group. Acceptability will be assessed by a six-question post-program questionnaire based on the barriers to engaging in physical activity. Questions relating to perceived importance and satisfaction with the program, any discomfort felt during training, difficulty of the exercises, appropriateness of duration and usefulness on daily activity will be asked to rate from a 5-point Likert scale from 'Strongly disagree' to 'Strongly agree', and be collected at the end of the intervention.
Frailty status | Baseline (Week 0) and Post-treatment (Week 10)
  Measured by the Tilburg frailty indicator (TFI).
  * There are 15 items in total, with a score of 0 or 1 on each item. The total score ranges from 0 to 15 points. A higher score mean a worse outcome (Higher frailty level).
  * A total score of >/=5 has a validity of 0.86 to determine the frailty status of the community-dwelling older Chinese population (Dong et al., 2017).
Frailty Status | Baseline (Week 0) and Post-treatment (Week 10)
  Measured by Fried Frailty Phenotype (FFP).
  * It consists of 5 components in assessing the severity of frailty, including weight loss, weakness, exhaustion, slowness and low physical activity, with a score of 0 or 1 for each component.
  * The total score ranges from 0 to 5 points. A higher score mean a worse outcome. The frailty status is categorized into robust (0), pre-frail (1-2), and frail (3-5).
Frailty status | Baseline (Week 0) and Post-treatment (Week 10)
  Measured by Short Physical Performance Battery (SPPB).
  * The SPPB is an assessment tool for participants' physical function and can be used to show the physical frailty.
  * It includes 3 components: standing balance, 4-m gait speed, and five-repetition sit-to-stand motion. Each component has a score of 0-4. The total score ranges from 0 to 12 points. A higher score mean a worse outcome.
  * A total score of <9 is regarded as frail.

SECONDARY OUTCOMES:
Cognitive function | Baseline (Week 0) and Post-treatment (Week 10)
  Measured by Hong Kong version Montreal Cognitive Assessment (HK-MoCA).
  * The score ranges from 0 to 30 points. A higher score indicates better cognitive function.
  * A score of 25 or below may indicate the presence of mild cognitive impairment.
Cognitive function | Baseline (Week 0) and Post-treatment (Week 10)
  Measured by forward digit span test.
  * Participants will be presented with a random series of digits and be asked to repeat them in the order presented.
  * A longer span indicates better working memory with high internal reliability.
Cognitive function | Baseline (Week 0) and Post-treatment (Week 10)
  Measured by Cognitive failures questionnaire (CFQ) (Chinese version), a self-report measure to assess individual forgetfulness, distractibility, and false triggering in everyday life.
  - It has 25 items (0-4 points). The total score ranges from 0 to 100 points. A higher point indicates fewer cognitive difficulties in daily life.
Pain level | Baseline (Week 0) and Post-treatment (Week 10)
  The average pain score will be assessed by the Numerical Pain Rating Scale (NPRS).
  * Participants will be asked to rate the average pain level on a scale from 0 (no pain) to 10 (maximal pain).
  * A higher score mean a worse outcome (higher pain level).
Health-related quality of life | Baseline (Week 0) and Post-treatment (Week 10)
  Measured by EuroQoL 5-Dimension 5-Level (EQ-5D-5L) (Hong Kong Chinese version) questionnaire.
  * The questionnaire consists of 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension will be rated from 1 (no problem) to 5 (extreme problems). A higher score mean a worse outcome.
  * It also has an EQ-VAS scale to self-rate the overall health perception from 0 (worst health) to 100 (best health). A higher score mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Yau, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- PolyU Institutional Review Board, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Only anonymised data will be shared to others when requested after publication is released. The anonymised data will be stored at the institutional data repository.

REFERENCES:
- [Background] Borg, G. (1998). Borg's Perceived Exertion and Pain Scales. Champaign, IL: Human Kinetics.
- [Background] Liguori, G., Feito, Y., Fountaine, C. (Charles J., & Roy, B. (Eds.). (2022). ACSM's guidelines for exercise testing and prescription (Eleventh edition.). Wolters Kluwer.
- [Background] Zhou, Y., Chen, J., Liu, Y., Wang, P., Zhu, L., & Yan, T. (2016). Validity and Reliability of the Cognitive Failures Questionnaire in Chinese College Students. Chinese Journal of Clinical Psychology, 24(3), 438-443.
- [Background] Frankenberg, C., Weiner, J., Knebel, M., Abulimiti, A., Toro, P., Herold, C. J., Schultz, T., & Schröder, J. (2021). Verbal fluency in normal aging and cognitive decline: Results of a longitudinal study. Computer Speech & Language, 68, 101195-. https://doi.org/10.1016/j.csl.2021.101195
- [Background] Winser S, Pang MYC, Rauszen JS, Chan AYY, Chen CH, Whitney SL. Does integrated cognitive and balance (dual-task) training improve balance and reduce falls risk in individuals with cerebellar ataxia? Med Hypotheses. 2019 May;126:149-153. doi: 10.1016/j.mehy.2019.03.001. Epub 2019 Mar 5. PMID 31010491
- [Background] Tiecker, A. P., Cadore, E. L., Izquierdo, M., Zmuda, G. G. O., Aguirre, F. B., & Bós, Â. J. G. (2024). Acceptability of a home-based multicomponent exercise program (Vivifrail®) for the oldest-old via videoconferencing during the Covid-19 pandemic. Revista Brasileira de Geriatria e Gerontologia., 27. https://doi.org/10.1590/1981-22562024027.230089.en
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Auyeung TW, Lee JS, Leung J, Kwok T, Woo J. The selection of a screening test for frailty identification in community-dwelling older adults. J Nutr Health Aging. 2014;18(2):199-203. doi: 10.1007/s12603-013-0365-4. PMID 24522474
- [Background] Wong EL, Cheung AW, Wong AY, Xu RH, Ramos-Goni JM, Rivero-Arias O. Normative Profile of Health-Related Quality of Life for Hong Kong General Population Using Preference-Based Instrument EQ-5D-5L. Value Health. 2019 Aug;22(8):916-924. doi: 10.1016/j.jval.2019.02.014. Epub 2019 Jul 27. PMID 31426933
- [Background] Wong A, Xiong YY, Kwan PW, Chan AY, Lam WW, Wang K, Chu WC, Nyenhuis DL, Nasreddine Z, Wong LK, Mok VC. The validity, reliability and clinical utility of the Hong Kong Montreal Cognitive Assessment (HK-MoCA) in patients with cerebral small vessel disease. Dement Geriatr Cogn Disord. 2009;28(1):81-7. doi: 10.1159/000232589. Epub 2009 Aug 11. PMID 19672065
- [Background] Varela-Vasquez LA, Minobes-Molina E, Jerez-Roig J. Dual-task exercises in older adults: A structured review of current literature. J Frailty Sarcopenia Falls. 2020 Jun 1;5(2):31-37. doi: 10.22540/JFSF-05-031. eCollection 2020 Jun. PMID 32510028
- [Background] Sugimoto T, Arai H, Sakurai T. An update on cognitive frailty: Its definition, impact, associated factors and underlying mechanisms, and interventions. Geriatr Gerontol Int. 2022 Feb;22(2):99-109. doi: 10.1111/ggi.14322. Epub 2021 Dec 9. PMID 34882939
- [Background] Simao R, Lemos A, Salles B, Leite T, Oliveira E, Rhea M, Reis VM. The influence of strength, flexibility, and simultaneous training on flexibility and strength gains. J Strength Cond Res. 2011 May;25(5):1333-8. doi: 10.1519/JSC.0b013e3181da85bf. PMID 21386731
- [Background] Salse-Batan J, Gonzalez-Devesa D, Dunabeitia I, Bidaurrazaga-Letona I, Ayan-Perez C, Sanchez-Lastra MA. Effects of stretching exercise on walking performance and balance in older adults: A systematic review and meta-analysis. Geriatr Nurs. 2025 Jan-Feb;61:479-490. doi: 10.1016/j.gerinurse.2024.12.018. Epub 2024 Dec 28. PMID 39733629
- [Background] Rast P, Zimprich D, Van Boxtel M, Jolles J. Factor structure and measurement invariance of the cognitive failures questionnaire across the adult life span. Assessment. 2009 Jun;16(2):145-58. doi: 10.1177/1073191108324440. Epub 2008 Dec 9. PMID 19066391
- [Background] Ramirez-Velez R, Lopez Saez de Asteasu M, Morley JE, Cano-Gutierrez CA, Izquierdo M. Performance of the Short Physical Performance Battery in Identifying the Frailty Phenotype and Predicting Geriatric Syndromes in Community-Dwelling Elderly. J Nutr Health Aging. 2021;25(2):209-217. doi: 10.1007/s12603-020-1484-3. PMID 33491036
- [Background] Perracini MR, Mello M, de Oliveira Maximo R, Bilton TL, Ferriolli E, Lustosa LP, da Silva Alexandre T. Diagnostic Accuracy of the Short Physical Performance Battery for Detecting Frailty in Older People. Phys Ther. 2020 Jan 23;100(1):90-98. doi: 10.1093/ptj/pzz154. PMID 31612228
- [Background] Pereira Oliva HN, Mansur Machado FS, Rodrigues VD, Leao LL, Monteiro-Junior RS. The effect of dual-task training on cognition of people with different clinical conditions: An overview of systematic reviews. IBRO Rep. 2020 Jul 1;9:24-31. doi: 10.1016/j.ibror.2020.06.005. eCollection 2020 Dec. PMID 33336101
- [Background] Pandey A, Kitzman D, Reeves G. Frailty Is Intertwined With Heart Failure: Mechanisms, Prevalence, Prognosis, Assessment, and Management. JACC Heart Fail. 2019 Dec;7(12):1001-1011. doi: 10.1016/j.jchf.2019.10.005. PMID 31779921
- [Background] Otones Reyes P, Garcia Perea E, Pedraz Marcos A. Chronic Pain and Frailty in Community-Dwelling Older Adults: A Systematic Review. Pain Manag Nurs. 2019 Aug;20(4):309-315. doi: 10.1016/j.pmn.2019.01.003. Epub 2019 May 16. PMID 31103515
- [Background] Negm AM, Kennedy CC, Thabane L, Veroniki AA, Adachi JD, Richardson J, Cameron ID, Giangregorio A, Petropoulou M, Alsaad SM, Alzahrani J, Maaz M, Ahmed MM, Kim E, Tehfe H, Dima R, Sabanayagam K, Hewston P, Abu Alrob H, Papaioannou A. Management of Frailty: A Systematic Review and Network Meta-analysis of Randomized Controlled Trials. J Am Med Dir Assoc. 2019 Oct;20(10):1190-1198. doi: 10.1016/j.jamda.2019.08.009. PMID 31564464
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Nascimbeni A, Caruso S, Salatino A, Carenza M, Rigano M, Raviolo A, Ricci R. Dual task-related gait changes in patients with mild cognitive impairment. Funct Neurol. 2015 Jan-Mar;30(1):59-65. PMID 26214028
- [Background] Matysiak O, Kroemeke A, Brzezicka A. Working Memory Capacity as a Predictor of Cognitive Training Efficacy in the Elderly Population. Front Aging Neurosci. 2019 May 31;11:126. doi: 10.3389/fnagi.2019.00126. eCollection 2019. PMID 31214015
- [Background] Macuco CR, Batistoni SS, Lopes A, Cachioni M, da Silva Falcao DV, Neri AL, Yassuda MS. Mini-Mental State Examination performance in frail, pre-frail, and non-frail community dwelling older adults in Ermelino Matarazzo, Sao Paulo, Brazil. Int Psychogeriatr. 2012 Nov;24(11):1725-31. doi: 10.1017/S1041610212000907. Epub 2012 Jun 1. PMID 22652040
- [Background] Gobbens RJ, van Assen MA, Luijkx KG, Wijnen-Sponselee MT, Schols JM. The Tilburg Frailty Indicator: psychometric properties. J Am Med Dir Assoc. 2010 Jun;11(5):344-55. doi: 10.1016/j.jamda.2009.11.003. Epub 2010 May 8. PMID 20511102
- [Background] Ghai S, Ghai I, Effenberg AO. Effects of dual tasks and dual-task training on postural stability: a systematic review and meta-analysis. Clin Interv Aging. 2017 Mar 23;12:557-577. doi: 10.2147/CIA.S125201. eCollection 2017. PMID 28356727
- [Background] Ferraz MB, Quaresma MR, Aquino LR, Atra E, Tugwell P, Goldsmith CH. Reliability of pain scales in the assessment of literate and illiterate patients with rheumatoid arthritis. J Rheumatol. 1990 Aug;17(8):1022-4. PMID 2213777
- [Background] Dong L, Liu N, Tian X, Qiao X, Gobbens RJJ, Kane RL, Wang C. Reliability and validity of the Tilburg Frailty Indicator (TFI) among Chinese community-dwelling older people. Arch Gerontol Geriatr. 2017 Nov;73:21-28. doi: 10.1016/j.archger.2017.07.001. Epub 2017 Jul 15. PMID 28734173
- [Background] Dent E, Lien C, Lim WS, Wong WC, Wong CH, Ng TP, Woo J, Dong B, de la Vega S, Hua Poi PJ, Kamaruzzaman SBB, Won C, Chen LK, Rockwood K, Arai H, Rodriguez-Manas L, Cao L, Cesari M, Chan P, Leung E, Landi F, Fried LP, Morley JE, Vellas B, Flicker L. The Asia-Pacific Clinical Practice Guidelines for the Management of Frailty. J Am Med Dir Assoc. 2017 Jul 1;18(7):564-575. doi: 10.1016/j.jamda.2017.04.018. PMID 28648901
- [Background] da Camara SM, Alvarado BE, Guralnik JM, Guerra RO, Maciel AC. Using the Short Physical Performance Battery to screen for frailty in young-old adults with distinct socioeconomic conditions. Geriatr Gerontol Int. 2013 Apr;13(2):421-8. doi: 10.1111/j.1447-0594.2012.00920.x. Epub 2012 Aug 6. PMID 22882512
- [Background] Daenen L, Varkey E, Kellmann M, Nijs J. Exercise, not to exercise, or how to exercise in patients with chronic pain? Applying science to practice. Clin J Pain. 2015 Feb;31(2):108-14. doi: 10.1097/AJP.0000000000000099. PMID 24662498
- [Background] Conway AR, Kane MJ, Bunting MF, Hambrick DZ, Wilhelm O, Engle RW. Working memory span tasks: A methodological review and user's guide. Psychon Bull Rev. 2005 Oct;12(5):769-86. doi: 10.3758/bf03196772. PMID 16523997
- [Background] Coelho-Junior HJ, Uchida MC. Effects of Low-Speed and High-Speed Resistance Training Programs on Frailty Status, Physical Performance, Cognitive Function, and Blood Pressure in Prefrail and Frail Older Adults. Front Med (Lausanne). 2021 Jul 26;8:702436. doi: 10.3389/fmed.2021.702436. eCollection 2021. PMID 34381802
- [Background] Chaplin WJ, McWilliams DF, Millar BS, Gladman JRF, Walsh DA. The bidirectional relationship between chronic joint pain and frailty: data from the Investigating Musculoskeletal Health and Wellbeing cohort. BMC Geriatr. 2023 May 5;23(1):273. doi: 10.1186/s12877-023-03949-4. PMID 37147635
- [Background] Cesari M, Calvani R, Marzetti E. Frailty in Older Persons. Clin Geriatr Med. 2017 Aug;33(3):293-303. doi: 10.1016/j.cger.2017.02.002. Epub 2017 Apr 6. PMID 28689563
- [Background] Castano LAA, Castillo de Lima V, Barbieri JF, de Lucena EGP, Gaspari AF, Arai H, Teixeira CVL, Coelho-Junior HJ, Uchida MC. Resistance Training Combined With Cognitive Training Increases Brain Derived Neurotrophic Factor and Improves Cognitive Function in Healthy Older Adults. Front Psychol. 2022 Oct 14;13:870561. doi: 10.3389/fpsyg.2022.870561. eCollection 2022. PMID 36312128
- [Background] Broadbent DE, Cooper PF, FitzGerald P, Parkes KR. The Cognitive Failures Questionnaire (CFQ) and its correlates. Br J Clin Psychol. 1982 Feb;21(1):1-16. doi: 10.1111/j.2044-8260.1982.tb01421.x. PMID 7126941
- [Background] Brigola AG, Rossetti ES, Dos Santos BR, Neri AL, Zazzetta MS, Inouye K, Pavarini SCI. Relationship between cognition and frailty in elderly: A systematic review. Dement Neuropsychol. 2015 Apr-Jun;9(2):110-119. doi: 10.1590/1980-57642015DN92000005. PMID 29213952
- [Background] Bridger RS, Johnsen SA, Brasher K. Psychometric properties of the Cognitive Failures Questionnaire. Ergonomics. 2013;56(10):1515-24. doi: 10.1080/00140139.2013.821172. Epub 2013 Jul 23. PMID 23879800
- [Background] Blyth FM, Noguchi N. Chronic musculoskeletal pain and its impact on older people. Best Pract Res Clin Rheumatol. 2017 Apr;31(2):160-168. doi: 10.1016/j.berh.2017.10.004. Epub 2017 Nov 4. PMID 29224694
- [Background] Alcon C, Bergman E, Humphrey J, Patel RM, Wang-Price S. The Relationship between Pain Catastrophizing and Cognitive Function in Chronic Musculoskeletal Pain: A Scoping Review. Pain Res Manag. 2023 Sep 9;2023:5851450. doi: 10.1155/2023/5851450. eCollection 2023. PMID 37719894
- See also: Izquierdo, M., Casas-Herrero, A., Zambom-Ferraresi, F., Martínez-Velilla, N., Alonso-Bouzón, C., & Rodriguez-Mañas, L. (2017). A practical guide for prescribing a multi-component physical training program to prevent weakness and falls in people over 70. — https://vivifrail.com/wp-content/uploads/2019/11/VIVIFRAIL-ENG-Interactivo.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT07035327/Prot_SAP_002.pdf